CLINICAL TRIAL: NCT00902044
Title: Administration of Her2 Chimeric Antigen Receptor Expressing T Cells for Subjects With Advanced Sarcoma (HEROS)
Brief Title: Her2 Chimeric Antigen Receptor Expressing T Cells in Advanced Sarcoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other); Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, Nabil Ahmed, Associate Professor, Pediatric Hematology Oncology, Center for Cell and Gene Therapy, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24489-HEROS; HEROS (Other: Baylor College of Medicine)
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Sarcoma
Keywords: Refractory Sarcoma; Metastatic Sarcoma; Sarcoma; HER2-positive; Gene Therapy; HER2-specific T cells
MeSH Terms: conditions — Sarcoma | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Autologous HER2-specific T cells (Experimental): THIS ARM IS CLOSED
  Dose Level 1: 1x10^4 cells/m2
  Dose Level 2: 3x10^4 cells/m2
  Dose Level 3: 1x10^5 cells/m2 (NOT BEING USED)
  Dose Level 4: 3x10^5 cells/m2 (NOT BEING USED)
  Dose Level 5: 1x10^6 cells/m2
  Dose Level 6: 3x10^6 cells/m2
  Dose Level 7: 1x10^7 cells/m2
  Dose Level 8: 3x10^7 cells/m2
  Dose Level 9: 1x10^8 cells/m2
  Interventions: Genetic: Autologous HER2-specific T cells
- HER2-specific T cells+fludarabine (Experimental): Autologous HER2-specific T cells+fludarabine:
  Dose Level 9A: fludarabine followed by 1x10^8 cells/m^2
  Interventions: Genetic: Autologous HER2-specific T cells; Drug: Fludarabine
- HER2-specific T cells+fludarab.+cycloph. (Experimental): Autologous HER2-specific T cells+fludarabine+cyclophosphamide:
  Dose Level 9B: fludarabine + cyclophosphamide followed by 1x10^8 cells/m^2
  Interventions: Genetic: Autologous HER2-specific T cells; Drug: Fludarabine; Drug: Cyclophosphamide
- CAR Positive cells (Experimental): Dose Level 9C: fludarabine + cyclophosphamide followed by 1x10^8 cells/m^2 CAR positive cells/m^2
  Interventions: Genetic: Autologous HER2-specific T cells; Drug: Fludarabine; Drug: Cyclophosphamide; Genetic: Autologous CAR Positive T cells

INTERVENTIONS:
Genetic: Autologous HER2-specific T cells — Each patient will receive one intravenous injection of autologous HER2-specific T cells at one of the dose levels. If the patient has stable disease or a reduction in the size of the tumor they can receive additional doses of HER2-specific T cells at 6 to 12 weeks intervals-each of which will consist of the same cell number as their HER2-specific T-cell injection. For the first two subsequent HER2-specific T-cell infusions, patients will be able to receive additional lymphodepleting chemotherapy according to their dose levels.
Drug: Fludarabine — Fludarabine will be administered for 5 days prior to the T cells
  The dose:
  >10 kg: 25 mg/m2/day;
  <10 kg: 1 mg/kg/day IV over 30 minutes
  Other Names: Fludara
  Arms: CAR Positive cells; HER2-specific T cells+fludarab.+cycloph.; HER2-specific T cells+fludarabine
Drug: Cyclophosphamide — Cyclophosphamide will be administered for 2 days.
  Fludarabine and cyclophosphamide will be given for 2 days, followed by fludarabine alone for the next 3 days, followed by 2 days of rest, before the T cells will be administered.
  Cyclophosphamide Dose:
  30 mg/kg/day IV over 1 hour (with Mesna and IV hydration)
  Fludarabine Dose:
  >10 kg: 25 mg/m2/day; <10 kg: 1 mg/kg/day IV over 30 minutes
  Other Names: Cytoxan
  Arms: CAR Positive cells; HER2-specific T cells+fludarab.+cycloph.
Genetic: Autologous CAR Positive T cells — Patient will receive one intravenous injection of autologous CAR T cells at dose level 9C. Further CAR T-cell dose escalation at dose level 9C will be done using the lymphodepletion schema as in dose level 9B.
  Arms: CAR Positive cells

SUMMARY:
Patients have a type of cancer called sarcoma. Because there is no standard treatment for the patients cancer at this time or because the currently used treatments do not work fully in all cases, patients are being asked to volunteer to take part in a gene transfer research study using special immune cells. This research study combines two different ways of fighting disease: antibodies and T cells. Antibodies are proteins that protect the body from diseases caused by germs or toxic substances. They work by binding those germs or substances, which stops them from growing or exerting their toxic effects. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including tumor cells or cells that are infected with germs. Both antibodies and T cells have been used to treat patients with cancers: they both have shown promise, but have not been strong enough to cure most patients. We have found from previous research that we can put a new gene into T cells that will make them recognize cancer cells and kill them. We now want to see if we can put a new gene in these cells that will let the T cells recognize and kill sarcoma cells. The new gene that we will put in makes an antibody specific for HER2 (Human Epidermal Growth Factor Receptor 2) that binds to sarcoma cells. In addition it contains CD28, which stimulated T cells and make them last longer. In other clinical studies using T cells, some investigators found that giving chemotherapy before the T cell infusion can improve the amount of time the T cells stay in the body and therefore the effect the T cells can have. Giving chemotherapy before a T cell infusion is called lymphodepletion since the chemotherapy is specifically chosen to decrease the number of lymphocytes in the body. Decreasing the number of patient's lymphocytes first should allow the T cells we infuse to expand and stay longer in your body, and potentially kill cancer cells more effectively. We will use fludarabine or the combination of cyclophosphamide and fludarabine as the chemotherapy agents for lymphodepletion. Cyclophosphamide and fludarabine are the chemotherapy agents most commonly used for lymphodepletion in immunotherapy clinical trials. The purpose of this study is to find the largest safe dose of chimeric T cells, and to see whether this therapy might help patients with sarcoma. Another purpose is to see if it is safe to give HER2-CD28 T cells after lymphodepleting chemotherapy.

DETAILED DESCRIPTION:
Because the cells have a new gene in them the patient will be followed for a total of 15 years to see if there are any long term side effects of gene transfer.

When the patient is enrolled on this study, they will be assigned a dose of HER2-CD28 T cells. Depending on which dose level they are assigned, they will receive one of the following:

HER2-CD28 T cells and fludarabine (patient will receive fludarabine for 5 days followed by injection of HER2-CD28 T cells)

OR

HER2-CD28 T cells, fludarabine and cyclophosphamide (patient will receive fludarabine and cyclophosphamide for 2 days, fludarabine alone for an additional 3 days, and 2 days of rest before receiving the HER2-CD28 T cells.).

The HER2-CD28 T cells will be given into the vein through an IV line. The injection will take between 1 and 10 minutes. The patient will be followed in the clinic after the injection for 1 to 4 hours.

Each patient will be followed for 6 weeks after the T-cell infusion for evaluation of toxicity. They will have standard tests and procedures as well as research blood draws.

If the patient has stable disease (the tumor did not grow) or there is a reduction in the size of the tumor on imaging studies after the T-cell infusion, they can receive additional doses of the T cells at 6 to 12 weeks intervals. For the first two subsequent HER2-specific T-cell infusions, patients will be able to receive additional lymphodepleting chemotherapy according to their dose levels.

ELIGIBILITY:
INCLUSION CRITERIA:

Procurement Eligibility:

1. Diagnosis of refractory HER2-positive sarcoma or metastatic HER2-positive osteosarcoma.
2. Karnofsky/Lansky score of 50 or greater
3. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

Treatment Eligibility:

1. Diagnosis of refractory HER2-positive sarcoma or metastatic HER2-positive sarcoma with disease progression after receiving at least one prior systemic therapy.
2. Recovered from acute toxic effects of all prior cytotoxic chemotherapy at least 4 weeks before entering this study. PD1/PDL1 inhibitors will be allowed to continue during treatment if medically indicated.
3. Normal ECHO (Left ventricular ejection fraction (LVEF) has to be within normal, institutional limits)
4. Life expectancy 6 weeks or greater
5. Karnofsky/Lansky score of 50 or greater
6. Bilirubin 3x or less, AST 3x or less, Serum creatinine 2x upper limit of normal or less, Hgb 7.0 g/dl or greater, WBC greater than 2,000/ul, ANC greater than 1,000/ul, platelets greater than 100,000/ul. Creatinine clearance is needed for patients with creatinine greater than 1.5 times upper limit of normal.
7. Pulse oximetry of 90% or greater on room air
8. Sexually active patients must be willing to utilize one of the more effective birth control methods for 6 months after the CTL infusion. Male partner should use a condom
9. Available autologous transduced T lymphocytes with 15% or more expression of HER2 CAR as determined by flow-cytometry and killing of HER2-positive targets 20 % or greater in cytotoxicity assay.
10. Chest radiograph for baseline evaluation of lungs
11. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent

EXCLUSION CRITERIA:

At time of Procurement:

1. Known HIV positivity
2. Severe previous toxicity from cyclophosphamide or fludarabine

At time of Treatment:

1. Severe intercurrent infection
2. Known HIV positivity
3. Pregnant or lactating
4. History of hypersensitivity reactions to murine protein-containing products
5. Severe previous toxicity from cyclophosphamide or fludarabine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2010-02-11; Primary Completion 2019-12-06 (Actual); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicity after one injection of HER2-specific T cells | 6 weeks
  To determine the safety of one intravenous injection of autologous T cells expressing HER2-specific chimeric antigen receptor (CAR) in patients with advanced HER2-positive sarcoma.
  To determine the safety of one intravenous injection of 1x10^8/m^2 autologous T cells after lymphodepleting chemotherapy.

SECONDARY OUTCOMES:
Frequency of HER2-specific T cells pre and post injection | 15 years
  To assess the in vivo expansion and persistence of infused T cells using immunoassays and transgene detection
Change in tumor size from pre to post injection | 6 weeks
  To assess the anti-tumor effects of the infused HER2-specific T cells

CONTACTS AND LOCATIONS:
Overall Officials: Nabil M Ahmed, MD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] Hegde M, Navai S, DeRenzo C, Joseph SK, Sanber K, Wu M, Gad AZ, Janeway KA, Campbell M, Mullikin D, Nawas Z, Robertson C, Mathew PR, Zhang H, Mehta B, Bhat RR, Major A, Shree A, Gerken C, Kalra M, Chakraborty R, Thakkar SG, Dakhova O, Salsman VS, Grilley B, Lapteva N, Gee A, Dotti G, Bao R, Salem AH, Wang T, Brenner MK, Heslop HE, Wels WS, Hicks MJ, Gottschalk S, Ahmed N. Autologous HER2-specific CAR T cells after lymphodepletion for advanced sarcoma: a phase 1 trial. Nat Cancer. 2024 Jun;5(6):880-894. doi: 10.1038/s43018-024-00749-6. Epub 2024 Apr 24. PMID 38658775
- [Derived] Hegde M, Joseph SK, Pashankar F, DeRenzo C, Sanber K, Navai S, Byrd TT, Hicks J, Xu ML, Gerken C, Kalra M, Robertson C, Zhang H, Shree A, Mehta B, Dakhova O, Salsman VS, Grilley B, Gee A, Dotti G, Heslop HE, Brenner MK, Wels WS, Gottschalk S, Ahmed N. Tumor response and endogenous immune reactivity after administration of HER2 CAR T cells in a child with metastatic rhabdomyosarcoma. Nat Commun. 2020 Jul 15;11(1):3549. doi: 10.1038/s41467-020-17175-8. PMID 32669548

DOCUMENTS (1):
  • Informed Consent Form (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT00902044/ICF_000.pdf